CLINICAL TRIAL: NCT01754961
Title: Effects of Vitamin D on Inflammation in Liver Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Veterans Medical Research Foundation (Other)
Responsible Party: Principal Investigator, Mario Chojkier, Professor of Medicine, Veterans Medical Research Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UCSD-111219
Record Dates: First submitted 2011-11-17; First posted 2012-12-21 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Hepatitis C Infection; Vitamin D Deficiency
MeSH Terms: conditions — Hepatitis C; Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo will be given on Day 1 orally
  Interventions: Drug: Placebo
- Vitamin D (Active Comparator): Administration of 500,000 IU Vitamin D orally on Day 1
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Vitamin D 500,000 IU given orally on Day 1
  Other Names: Vitamin D Drug
  Arms: Vitamin D
Drug: Placebo — Placebo given orally on Day 1
  Other Names: Emulsion placebo
  Arms: Placebo

SUMMARY:
Chronic liver diseases are associated with inflammation. The investigators postulate that Vitamin D may modulate inflammation. Thus the investigators will study the effect of Vitamin D replacement in patients with Hepatitis C infection and Vitamin D deficiency.

DETAILED DESCRIPTION:
Vitamin D appears to be a critical signaling molecule for macrophages because is needed for activation and differentiation of monocytes/macrophages. From our Preliminary Studies( VA Merit Review Grant), we propose that Vitamin D deficiency may alter the 'pro-inflammatory' ('classically activated') M1 macrophages , characterized by i] high expression of NOS2, TNF-a, IL-1, IL-6, IL-8, TGF-a, CXCL10, and CCL19; and ii] minimal expression of arginase 1 and mannose R.

The clinical relevance of these findings is suggested by the presence of activated M1 macrophages in liver biopsies from patients with severe drug-induced liver injury (unpublished observations).

Prospective vitamin D supplementation studies with appropriate endpoints are needed to define the role of vitamin D on inflammation in patients with chronic liver diseases.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 or older
* Total 25-OH Vit D < 25 ng/mL
* Infection with HCV genotype 1 (subjects infected with multiple genotypes are not eligible).
* Plasma HCV RNA concentration of >100,000 IU/mL.
* HCV-infected subjects naïve to treatment: subjects who either have never been treated for HCV infection or who previously received HCV treatment ending > 3 months prior to enrollment (including, any IFN-Alpha with or without ribavirin, or other anti-HCV antiviral medication).

Exclusion Criteria:

* Women who are pregnant or breastfeeding.
* Patients with Sarcoidosis, Histoplasmosis, Lymphoma, Primary Hyperparathyroidism or Idiophatic Hypercalcemia.
* Liver Cirrhosis.
* Known active gastrointestinal disease that could interfere with the absorption of the test article.
* Laboratory determinations at screening as follows:
* Hemoglobin <10 g/dL .
* Serum creatinine that is not within normal limits. However, such subjects may be enrolled if the Cockroft-Gault glomerular filtration rate (GFR) is > 50 mL/minute.
* Unstable hypertension, cardiac disease or type 2 diabetes requiring changes in treatment with medications 4 weeks prior to screening or during the screening period.
* Use of an investigational drug within 4 weeks before the screening visit or during the screening period.
* Use of systemic immunosuppressants (including systemic, oral, or intravenous corticosteroids) or immunomodulating agents within 4 weeks before the screening visit or during the screening period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-10 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Macrophage activation | one week
  As determined by serum levels and macrophage cytokine production compared to placebo and baseline

SECONDARY OUTCOMES:
Liver injury | one week
  Measurement of ALT/AST

CONTACTS AND LOCATIONS:
Overall Officials: Mario Chojkier, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UC San Diego, CTRI, La Jolla, California, United States